

## Moorfields Eye Hospital NHS Foundation Trust

City Road London EC1V 2PD

Tel: 020 7253 3411 www.moorfields.nhs.uk

Full title of trial Prospective non-randomised exploratory

study to assess the safety and efficacy of

Eylea in cystoid macular oedema associated with Retinitis Pigmentosa

Short title Aflibercept for Macular Oedema with

Underlying Retinitis Pigmentosa (AMOUR)

study

**Version and date of consent form:** Version 1.1 14<sup>th</sup> March 2016

**Sponsor:** Moorfields Eye Hospital NHS Foundation

Trust

Sponsor protocol number MICM1014

Funder (s): Bayer PLC

**EudraCT no** 2015-003723-65

ACTIVE IMP(s): Aflibercept (Eylea)

PLACEBO IMP(s): N/A

Phase of trial Therapeutic exploratory trial (phase II)

Sites(s) Single site – Moorfields Eye Hospital

## **Chief investigator:**

Professor Michel Michaelides Moorfields Eye Hospital City Road London EC1V 2PD UK

Department of Genetics
UCL Institute of Ophthalmology
11-43 Bath Street
London
EC1V 9EL
UK

## **Sponsor Representative:**

Gisela Barreto
Research Portfolio Manager
Moorfields Eye Hospital NHS Foundation
Trust
162 City Road
London
EC1V 2PD

## **CONSENT FORM**

**Study Title:** Aflibercept for Macular Oedema with Underlying Retinitis Pigmentosa (AMOUR) trial

| Patient ID: | |
|---|---|
| <b>Researchers:</b> Dr. Stacey Strong, Professor Michel Michaelides, and Professor Awebster | Andrew |
| Please initia | l box |
| <ol> <li>I confirm that I have read and understand the information sheet dated<br/>version 2.1 dated 14<sup>th</sup> March 2016 for the above study and have had<br/>the opportunity to ask questions.</li> </ol> | |
| <ol> <li>I understand that my participation is voluntary and that I am free to<br/>withdraw at any time, without giving any reason and without my<br/>medical care or legal rights being affected.</li> </ol> | |
| <ol> <li>I understand that sections of my medical notes may be looked<br/>at by responsible individuals from Moorfields Eye Hospital or from<br/>regulatory authorities where it is relevant to my taking part in research.<br/>I give permission for these individuals to have access to my records.</li> </ol> | |
| <ol> <li>I understand that my GP will be informed of my participation in this<br/>research project and of any findings significant to my general health</li> </ol> | |
| 5. I understand that I will not benefit financially from participating in the study | |
| 6. I agree to take part in the above study. | |
| For women of child bearing potential only | |
| 7. I understand that if I am a woman of child bearing potential I will be asked to undertake a pregnancy test prior to enrolment. I agree to use adequate contraception throughout the duration of the trial (12 months) and for at least 3 months after my last injection. I agree to be monitored | |

by my GP +/- obstetrics and gynaecology team should I fall pregnant during my participation in the study or within 3 months of my last

injection.

| Name of patient | Date | Signature |
|---|---|---|
| Name of person taking consent (if different from researcher) | Date | Signature |
| Researcher | <br>Date | Signature |

When completed: Original for researcher site file; a copy for the participant; a copy for the medical notes.